CLINICAL TRIAL: NCT05261048
Title: Effects of Pelvic Proprioceptive Neuromuscular Facilitation on Trunk Control and Balance in Children With Spastic Hemiplegic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Pelvic Proprioceptive Neuromuscular Facilitation on Trunk Control and Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/1073/2021
Record Dates: First submitted 2022-02-12; First posted 2022-03-02 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: Unilateral cerebral palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcome Assessor) Study will be single blinded. The assessor will be unaware of the treatment given to both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Proprioceptive neuromuscular facilitation in addition to Conventional Physical Therapy (Experimental): The experimental group received both conventional and Pelvic PNF for 30 minutes each, once in a day, 4 days per week.
  The experimental group will be given anterior elevation-Posterior depression pattern with the techniques of Rhythmic initiation, Slow reversal and Stabilizing reversal.
  These techniques will be given on affected side for total 30 minutes with 15 minutes of pelvic PNF in one session with rest periods in between.
  Participants will be positioned into side lying with both hip flexion 1000 and knee flexion 450, neck supported by a pillow with flexion of 300.
  Hand placement for anterior elevation over the crest of the ilium one hand overlaps other for posterior depression heel of the one hand hold with other hand on the ischial tuberosity.
  "Pull up" and "Push down" command will be given along with the techniques of rhythmic initiation, slow reversal and stabilizing reversal.
  Interventions: Other: Pelvic Proprioceptive neuromuscular facilitation in addition to Conventional Physical Therapy; Other: Conventional Physical Therapy
- Conventional Physical Therapy (Placebo Comparator): Patient will perform conventional physiotherapy in form of truncal exercises, which consist of upper and lower part of trunk in spine and sitting position for total 30 minutes and then participants will be asked to take some rest. In supine position, pelvic bridging, unilateral pelvic bridging, upper trunk rotation (clasped hand), lower trunk rotation (crook lying) with 3 repetitions for each exercise.
  In sitting position, exercises included flexion and extension of lower trunk, rotation of upper and lower trunk, forward and lateral reach with 3 repetitions for each exercise.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Pelvic Proprioceptive neuromuscular facilitation in addition to Conventional Physical Therapy — The experimental group received both conventional and Pelvic PNF for 30 minutes each, once in a day, 4 days per week. The experimental group will be given anterior elevation-Posterior depression pattern with the techniques of Rhythmic initiation, Slow reversal and Stabilizing reversal. These techniques will be given on affected side for total 30 minutes with 15 minutes of pelvic PNF in one session with rest periods in between. Participants will be positioned into side lying with both hip flexion 1000 and knee flexion 450, neck supported by a pillow with flexion of 300. Hand placement for anterior elevation over the crest of the ilium one hand overlaps other for posterior depression heel of the one hand hold with other hand on the ischial tuberosity.
  "Pull up" and "Push down" command will be given along with the techniques of rhythmic initiation, slow reversal and stabilizing reversal.
  Arms: Pelvic Proprioceptive neuromuscular facilitation in addition to Conventional Physical Therapy
Other: Conventional Physical Therapy — Conventional physiotherapy will be asked to perform truncal exercises in spine and sitting position for total 30 minutes including rest periods in between, once in a day for 4 days per week.
  Exercises in supine position included (pelvic bridging, unilateral pelvic bridging, upper trunk rotation (clasped hand), lower trunk rotation (crook lying) with 3 repetitions for each exercise.
  In sitting position, exercises included flexion and extension of lower trunk, rotation of upper and lower trunk, forward and lateral reach with 3 repetitions for each exercise.

SUMMARY:
The study will be randomized controlled trial. This study will be conducted in Children Hospital Pakistan. A sample size of 60 will be randomly allocated into two groups, (30 participants in each group), by lottery method.

* The participants randomly allocated into control group A, will receive conventional physiotherapy in the form of truncal exercises, which consists of upper and lower part of the trunk in spine and sitting position for a total 30 minutes including rest periods in between, once in a day for 4 days per week.
* Participants in experimental group B receive both conventional physiotherapy and Pelvic Proprioceptive Neuromuscular Facilitation for 30 minutes, once in a day, 4 days per week for 12 weeks.
* The experimental group received anterior elevation-Posterior depression pattern with the techniques of Rhythmic initiation, Slow reversal and Stabilizing reversal.
* Affected side of the pelvis was given these techniques for total 30 minutes with 15 minutes of pelvic PNF in one session with rest periods in between.
* Baseline data will be collected at baseline, 6 weeks and 12 weeks during follow up through Trunk Impairment scale (TIS) and Pediatric balance scale (PBS).

DETAILED DESCRIPTION:
* Recruitment: Participants who met the inclusion/exclusion will be recruited from the outpatient Department of Pediatric Rehabilitation of the children hospital.
* Screening: Participants will be considered eligible for entering the study with Gross motor function level 1 and 2 ( walk with or without limitation) and spasticity range between grade 1 and 2 according Modified Ashworth scale.
* Gross Motor Function Classification System (GMFCS): Children who can walk independently without assistance are categorized into GMFCS levels I and II, whereas those who cannot walk independently and need assistance or gait assistive device for ambulation are categorized into levels III and V.
* Modified Ashworth scale: It will be assessed while moving from extension to flexion scoring 0 No increase in tone. 1 slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension. 1+ slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM). 2 more marked increase in tone but more marked increased in muscle tone through most limb easily flexed. 3 considerable increase in tone, passive movement difficult. 4 limb rigid in flexion or extension
* Randomization and allocation: Afterwards, participants will be conforming the eligibility criteria will be randomly allocated, through lottery method, into two experimental groups (Group A, Group B).
* Blindness: The study will be single blinded. The assessor will be unaware of the treatment given to both groups.
* Intervention: The participants randomly allocated to control group A, will receive conventional physical therapy in the form of truncal exercises, which consists of upper and lower part of the trunk in spine and sitting position for 30 minutes including rest intervals in between.
* Participants in experimental group B, will receive pelvic proprioceptive neuromuscular facilitation in addition to conventional physical therapy for 30 minutes each, once in a day, 4 days per week for 12 weeks.
* Duration: Forty eight sessions will be given over a period of 12 weeks for each session of 30 minutes.
* Outcome Variables and measures:

  1. Trunk Control(Trunk Impairment scale (TIS)
  2. Balance (Pediatric balance scale (PBS)
* Outcome measures will be taken at baseline, 6 weeks and 12 weeks during follow up.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as Spastic hemiplegic cerebral palsy
* Age group (5-12) years
* Both male and female
* Gross motor function level 1 and 2 ( walk with or without limitation)
* Spasticity range between grade 1 and 2 according Modified Ashworth scale
* Able to follow the simple verbal instructions.

Exclusion Criteria:

* Children with visual, auditory, vestibular or perceptual deficit.
* Any Fracture
* Other neurological and cardio logical conditions( mental disorder, epilepsy, autism)
* Cognitive impairments
* Other types of CP

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-11 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale | 12 weeks
  It is used to assess trunk control including static and dynamic-sitting balance, and upper and lower trunk coordination during trunk rotation while sitting. Each item was graded on a 2-4-point ordinal scale. The highest possible scores for the static- and dynamic-sitting balance tests, and the trunk coordination test were 7, 10, and 6, and the total TIS score ranged from 0 to 23. Each item of the TIS was tested three times and the highest score counted. No practice was allowed.

SECONDARY OUTCOMES:
Pediatric Balance Scale | 12 weeks
  Pediatric Balance Scale that is a modified version of the Berg Balance Scale. It is used to assess functional balance skills in school-aged children, from typically developing children and children with motor impairments. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.

CONTACTS AND LOCATIONS:
Overall Officials: Saiqa Irum, MS PTN, Principal Investigator — University of Lahore
Locations (1):
- Children Hospital, Faisalabad, Punjab/Muslim, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Background] Panibatla S, Kumar V, Narayan A. Relationship Between Trunk Control and Balance in Children with Spastic Cerebral Palsy: A Cross-Sectional Study. J Clin Diagn Res. 2017 Sep;11(9):YC05-YC08. doi: 10.7860/JCDR/2017/28388.10649. Epub 2017 Sep 1. PMID 29207820
- [Background] Upadhyay J, Tiwari N, Ansari MN. Cerebral palsy: Aetiology, pathophysiology and therapeutic interventions. Clin Exp Pharmacol Physiol. 2020 Dec;47(12):1891-1901. doi: 10.1111/1440-1681.13379. Epub 2020 Aug 19. PMID 32662125
- [Background] Sharma V, Kaur J. Effect of core strengthening with pelvic proprioceptive neuromuscular facilitation on trunk, balance, gait, and function in chronic stroke. J Exerc Rehabil. 2017 Apr 30;13(2):200-205. doi: 10.12965/jer.1734892.446. eCollection 2017 Apr. PMID 28503533
- [Background] Stepien A, Fabian K, Graff K, Podgurniak M, Wit A. An immediate effect of PNF specific mobilization on the angle of trunk rotation and the Trunk-Pelvis-Hip Angle range of motion in adolescent girls with double idiopathic scoliosis-a pilot study. Scoliosis Spinal Disord. 2017 Sep 6;12:29. doi: 10.1186/s13013-017-0132-0. eCollection 2017. PMID 28905003
- [Background] Kallem Seyyar G, Aras B, Aras O. Trunk control and functionality in children with spastic cerebral palsy. Dev Neurorehabil. 2019 Feb;22(2):120-125. doi: 10.1080/17518423.2018.1460879. Epub 2018 Apr 13. PMID 29652201
- [Background] Kim DH, An DH, Yoo WG. Changes in trunk sway and impairment during sitting and standing in children with cerebral palsy. Technol Health Care. 2018;26(5):761-768. doi: 10.3233/THC-181301. PMID 29991150
- [Background] Blair E. Epidemiology of the cerebral palsies. Orthop Clin North Am. 2010 Oct;41(4):441-55. doi: 10.1016/j.ocl.2010.06.004. PMID 20868877